CLINICAL TRIAL: NCT04155541
Title: Special Investigation for Vizimpro Tablets
Brief Title: Special Investigation for VIZIMPRO Tablets (Secondary Data Collection Study; Safety and Efficacy of VIZIMPRO Under Japanese Medical Practice)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7471048
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: EGFR Mutation-positive Inoperable or Reccrent NSCLC
Keywords: VIZIMPRO; EGFR mutation-positive inoperable or recurrent NSCLC; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VIZIMPRO(dacomitinib hydrate): Patients with EGFR mutation-positive inoperable or recorrent NSCLN (non-small cell lung cancer) who have not received VIZIMPRO (dacomitinib hydrate)
  Interventions: Drug: dacomitinib hydrate

INTERVENTIONS:
Drug: dacomitinib hydrate — The usual adult starting dosage for oral use is 45mg of dacomitinib hydrate once daily. The dose should be reduced appropriately according to the patient's condition.
  Other Names: VIZIMPRO

SUMMARY:
Secondary data collection study: safety and efficacy of VIZIMPRO under Japanese medical practice

ELIGIBILITY:
Inclusion Criteria:

* patient with EGFR mutation-positive inoprable or recurrent NSCLC who have not received VIZIMPRO(dacomitinib hydrate)

Exclusion Criteria:

* Exclusion criteria is not provided in this study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient who meet the inclusion criteria and who were registered to this study within 84 days including the start date of treatment with this product will be subjects for this study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
The number and proportion of patients with ILD (interstitial lung disease) | 52 weeks form the start date
  The number and proportion of patients with ILD (interstitial lung disease) will be tabulated by subgroup by risk factor

SECONDARY OUTCOMES:
Response rate | 52 weeks from the start date
  Response rate will be calculated. The response rate is defined as the propotion of patients with a best ovarall response of CR ro PR in the effectiveness analysis set.
The number and population of patients with adverse reactions | 52 weeks from the start date
  The number and population of patients with adverse reactions will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Japan, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471048